CLINICAL TRIAL: NCT06831370
Title: A Multicenter, Single-arm, Open-label, Phase 4 Study to Evaluate the Safety and Efficacy of Brentuximab Vedotin Plus Doxorubicin, Vinblastine and Dacarbazine in Indian Patients With Untreated Stage 3/4 Classical Hodgkin Lymphoma
Brief Title: A Study of Brentuximab Vedotin With Doxorubicin, Vinblastine and Dacarbazine in Adults With Hodgkin Lymphoma in India
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C25030
Record Dates: First submitted 2025-02-14; First posted 2025-02-18 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Hodgkin Lymphoma
Keywords: Lymphoma; Chemotherapy
MeSH Terms: conditions — Hodgkin Disease; Lymphoma | interventions — Brentuximab Vedotin; Doxorubicin; Vinblastine; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brentuximab Vedotin 1.2 mg/kg (Experimental): Participants will receive 1.2 milligrams per kilogram (mg/kg) brentuximab vedotin intravenous (IV) infusion on Days 1 and 15 of each 28-day cycle, within 1 hour after completion of treatment with other agents [25 milligrams per meter square (mg/m^2) doxorubicin, 6 mg/m^2 vinblastine and 375 mg/m^2 dacarbazine IV infusions] for a maximum of 6 cycles.
  Interventions: Drug: Brentuximab Vedotin; Drug: Doxorubicin; Drug: Vinblastine; Drug: Dacarbazine

INTERVENTIONS:
Drug: Brentuximab Vedotin — Brentuximab Vedotin IV infusion
  Other Names: Adcetris
Drug: Doxorubicin — Doxorubicin IV infusion
  Other Names: Adriamycin
Drug: Vinblastine — Vinblastine IV infusion
Drug: Dacarbazine — Dacarbazine IV infusion

SUMMARY:
The main aim of this study is to check how safe brentuximab vedotin is in adults with untreated Hodgkin Lymphoma (HL) when given together with doxorubicin (Adriamycin), vinblastine and dacarbazine therapy ('AVD'). Another aim is to learn how well treatment of brentuximab vedotin plus AVD works.

All participants will receive brentuximab vedotin plus AVD for approximately 6 months. Participants will undergo tests like Echocardiography (ECHO) and pulmonary function testing (PFT) during the study. ECHO is a test that uses ultrasound to show how the heart muscle and valves are working; PFT is a test to check how well a participant's lungs work.

Each participant will undergo a final health status check 2 months after the last treatment with brentuximab vedotin plus AVD.

ELIGIBILITY:
Inclusion Criteria

1. Treatment-naïve, Hodgkin lymphoma (HL) participants with Ann Arbor Stage 3 or 4 disease.

   Note: Participants must have histologically confirmed classical HL according to the current world health organization classification.
2. Participants must have bidimensional measurable disease as documented by radiographic technique (spiral computed tomography [CT] preferred) per the international working group revised criteria for response assessment for malignant lymphoma.
3. Male or female participants 18 years or older.
4. Eastern cooperative oncology group (ECOG) performance status less than or equal to (≤)2.
5. Female participants who:

   * Are postmenopausal for at least 1 year before the screening visit, OR
   * Are surgically sterile, OR
   * If they are of childbearing potential, agree to practice 1 highly effective method and 1 additional effective (barrier) method of contraception at the same time, from the time of signing of the informed consent form (ICF) through 6 months after the last dose of study drug, OR
   * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together).
6. Male participants, even if surgically sterilized (i.e., status post-vasectomy), who:

   * Agree to practice effective barrier contraception during the entire study treatment period and through 6 months after the last dose of study drug, OR
   * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods for the female partner], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together).
7. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.
8. Clinical laboratory values as specified below within 7 days before the first dose of study drug:

   * Absolute neutrophil count greater than or equal to (≥)1,000 per microliter (1,000/μL) unless there is known HL marrow involvement
   * Platelet count ≥75,000/μL unless there is known HL marrow involvement
   * Total bilirubin must be lesser than (<)1.5 x upper limit of the normal range (ULN) unless the elevation is known to be due to Gilbert syndrome.
   * Alanine Aminotransferase (ALT) or aspartate aminotransferase (AST) must be <3.0 x ULN. An AST and ALT may be elevated up to 5 times the ULN if their elevation can be reasonably ascribed to the presence of HL in liver.

Note: Moderate or severe hepatic disease patients will be excluded based upon Child-Pugh criteria.

* Serum creatinine must be <2.0 milligrams per deciliter (mg/dL) and/or creatinine clearance or calculated creatinine clearance >30 mL/minute (Cockcroft-Gault Equation).
* Hemoglobin must be ≥8 grams per deciliter (g/dL).

Exclusion Criteria

1. Female participants who are both lactating and breastfeeding or who have a positive serum pregnancy test during the screening period or a positive pregnancy test on Day 1 before first dose of study drug.
2. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
3. Known cerebral or meningeal disease (HL or any other etiology), including signs or symptoms of progressive multifocal leukoencephalopathy (PML).
4. Symptomatic neurologic disease compromising normal activities of daily living or requiring medications.
5. Any sensory or motor peripheral neuropathy.
6. Any active systemic viral, bacterial, or fungal infection requiring systemic antibiotics within 2 weeks prior to first study drug dose.
7. Prior immunosuppressive chemotherapy, therapeutic radiation, or any immunotherapy (e.g., immunoglobulin replacement, other monoclonal antibody therapies) within 12 weeks of first study drug dose.
8. Previously treated with brentuximab vedotin.
9. Any contraindications to the concomitant chemotherapy regimens (doxorubicin, vinblastine, and dacarbazine).
10. Known hypersensitivity to recombinant proteins, murine proteins, or to any excipient contained in the drug formulation of brentuximab vedotin or any component of doxorubicin, vinblastine, and dacarbazine (AVD).
11. Known human immunodeficiency virus (HIV) positive.
12. Known hepatitis B surface antigen-positive, or known or suspected active hepatitis C infection.
13. Diagnosed or treated for another malignancy within 3 years before the first dose or previously diagnosed with another malignancy and have any evidence of residual disease. Participants with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
14. Any of the following cardiovascular conditions or values within 6 months before the first dose of study drug:

    1. A left-ventricular ejection fraction <50%
    2. Myocardial infarction within 2 years of enrollment
    3. New York Heart Association (NYHA) Class 3 or 4 heart failure. Evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure (CHF), angina, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Adverse Drug Reactions (ADRs), and Unexpected ADRs | Up to 40 weeks
  An AE is defined as any untoward medical occurrence in a clinical investigation patient administered a drug; it does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. An SAE is any AE that results in death, is life-threatening, requires inpatient hospitalization or prolongation of an existing hospitalization, results in significant disability or incapacity, is a congenital anomaly/birth defect or is a medically important event. ADRs are defined as AEs which are in the investigator's opinion of causal relationship to the study treatment. An unexpected ADR is an ADR with the nature, severity, or outcome which is not consistent with summary of product characteristics.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Complete Remission (CR) | Up to 35 weeks
  CR is defined as disappearance of all the evidence of disease assessed by investigator per Revised Response Criteria for Malignant Lymphoma.
Objective Response Rate (ORR) | Up to 35 weeks
  ORR is defined as the disappearance of all evidences of a disease along with a decrease in evidences of a disease (CR+ partial remission [PR]) assessed by investigator per Revised Response Criteria for Malignant Lymphoma.
Positron Emission Tomography (PET) Negativity Rate at Cycle 2 | Days 20 to 28 of Cycle 2 (cycle length=28 days)
  The rate of PET negativity is the percentage of participants with PET negativity (defined as Deauville score 1, 2, or 3) at the end of Cycle 2. The Deauville 5-point scoring system is a five-point scoring system for the fluorodeoxyglucose (FDG) avidity of a Hodgkin's lymphoma or non-Hodgkin's lymphoma tumor mass as seen on FDG PET scan: Score 1= No uptake above the background, Score 2= Uptake ≤ mediastinum, Score 3= Uptake > mediastinum but ≤ liver, Score 4= Uptake moderately increased compared to the liver at any site, Score 5= Uptake markedly increased compared to the liver at any site or new lesions, Score X= New areas of uptake unlikely to be related to lymphoma. In this study, scores of 1, 2, and 3 are considered to be negative and scores of 4 and 5 are considered to be positive.
Progression Free Survival (PFS) | Up to 40 weeks
  PFS is defined as the time from study drug assignment to disease progression (PD) or death from any cause or date of last tumor assessment if the participant did not progress or die.
Overall Survival (OS) | Up to 40 weeks
  OS is defined as the time from study drug assignment to death from any cause or last date when the participant was known to be alive.
Disease Free Survival | Up to 40 weeks
  Disease free survival is measured from the time of occurrence of disease-free state or attainment of a CR to disease recurrence or death as a result of lymphoma or acute toxicity of treatment.
Event Free Survival | Up to 40 weeks
  Event free survival (time to treatment failure) is measured from the time from study entry to any treatment failure including disease progression, or discontinuation of treatment for any reason.
Duration of Response (DOR) | Up to 40 weeks
  DOR is defined as the time from first occurrence of overall response (CR or PR whichever is recorded first) after start of study treatment until the date of disease progression or relapse.
Duration of Complete Remission (DOCR) | Up to 40 weeks
  DOCR in participants with confirmed CR is the time between first documentation of CR and PD.

CONTACTS AND LOCATIONS:
Locations (11):
- India (11):
  - HCG City Cancer Centre, Vijayawada, Andhra Pradesh
  - Gauhati Medical college and Hospital, Guwahati, Assam
  - Unique Hospital Multispeciality and Research Institute, Surat, Gujarat
  - HCG Cancer Centre, Bangalore, Karnataka
  - JIPMER, Puducherry, Kerala
  - HCG Manavata Cancer Centre, Nashik, Maharashtra
  - ACTREC, Navi Mumbai, Maharashtra
  - DMH, Pune, Maharashtra
  - Rajiv Gandhi Cancer Hospital, Delhi, New Delhi
  - NRS Medical college & Hospital, Kolkata, Kolkata, West Bengal
  - AIIMS, New Delhi

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/9f6a2df9fa654e93??page=1&idFilter=C25030